CLINICAL TRIAL: NCT04774497
Title: Effect of Oxygen Inhalation on Fatigue After Chemotherapy of Breast Cancer in High Altitude Area
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiuda Zhao (Other)
Responsible Party: Sponsor-Investigator, Jiuda Zhao, Professor, Affiliated Hospital of Qinghai University
Organization: Affiliated Hospital of Qinghai University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AHQU-2021001
Record Dates: First submitted 2021-02-18; First posted 2021-03-01 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Chemotherapy; Fatigue; Oxygen; High altitude
MeSH Terms: conditions — Breast Neoplasms; Fatigue; Altitude Sickness | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxygen inhalation treatment group (Experimental): 1. Patients receive chemotherapy for breast cancer.
  2. Patients are randomly divided into inhalation treatment group. Oxygen inhalation is started on the first day of chemotherapy, and the oxygen inhalation volume is 2 L / min, 8 hours / day for 3 consecutive days.（d1，d2，d3）.
  3. Blood samples are collected before and after chemotherapy（d0，d3）.
  4. CIS and BFI are measured before chemotherapy（d0, d3 chemotherapy regimen/ d0, d3， chemotherapy regimen）.
  Interventions: Other: Oxygen inhalation treatment group
- Oxygen non-inhalation treatment group (Placebo Comparator): 1. Patients receive chemotherapy for breast cancer.
  2. Patients are randomly divided into non-inhalation treatment group.
  3. Blood samples are collected before and after chemotherapy（d0，d3）.
  4. CIS and BFI are measured before chemotherapy（d0, d3，chemotherapy regimen/ d0, d3， chemotherapy regimen）.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Oxygen inhalation treatment group — Oxygen inhalation group: oxygen inhalation was started on the first day of chemotherapy, and the oxygen inhalation volume was 2 L / min, 8 hours / day for 3 consecutive days.
  Arms: Oxygen inhalation treatment group
Other: Control group — The control group was not given oxygen inhalation.
  Arms: Oxygen non-inhalation treatment group

SUMMARY:
At present, there are few studies on the side effects of chemotherapy in breast cancer patients at high altitude area, and there are no studies on the relationship between oxygen inhalation and fatigue after chemotherapy in breast cancer patients at high altitude. The investigators intend to explore whether oxygen inhalation can improve fatigue at high altitude through this prospective randomized study. In our study, a single center, open-label, randomized phase 2 clinical trial will conduct to investigate whether oxygen inhalation during chemotherapy can improve chemotherapy-related fatigue in patients with breast cancer. The effects of oxygen inhalation on side effects of chemotherapy such as Cancer related fatigue (CRF) were observed. The investigators intend to explore whether oxygen therapy can improve fatigue at high altitude through this prospective randomized study. The investigators enrolled breast cancer patients before chemotherapy. The investigators will use the checklist individual strength(CIS) and the brief fatigue inventory (BFI) to evaluate the fatigue status of patients, and extract the blood of patients for evaluate blood pro-inflammatory cytokines IL-1 β, IL-6, C-reactive protein (CRP), transforming growth factor (TGF-β), soluble tumor necrosis factor (TNF) receptor II (sTNF-RII), inducible factor-1(HIF-1), Hypoxia inducible factor-2(HIF-2)in the plasma.

DETAILED DESCRIPTION:
Fatigue is the most common symptom experienced by patients from cancer diagnosis to the end of life. CRF is different from other types of fatigue. It is severe, persistent and can not be alleviated by rest or sleep. CRF affects nearly 65% of cancer patients, more than two-thirds believe that severe CRF lasts at least 6 months, and one-third report that fatigue persists for several years after chemotherapy.

The etiology of CRF has not been fully elucidated, although it may involve several physiological and biochemical systems, which may vary with tumor type, disease stage and treatment. Recently, several cytokines and other proinflammatory mediators produced in tryptophan degradation and cancer response are associated with fatigue; however, their direct role in the pathogenesis of fatigue remains controversial. Cytokines may play a role at a variety of levels, including mood, muscle mass, strength and metabolic status, and thus are associated with the pathophysiology of fatigue. Recent studies have shown that fatigue is positively correlated with circulating levels of inflammatory markers, especially IL-6, IL-1 and neopterin, which are significantly correlated with CRF. CRF is also common in breast cancer patients, and the incidence rate of CRF is increasing as the incidence of breast cancer increases. In the treatment of breast cancer patients， chemotherapy can cause some patients' non hematological side effects such as fatigue. During the chemotherapy of breast cancer at high altitude area, clinical observation showed that the incidence rate of side effects after chemotherapy was higher in plateau area. Retrospectively analyzed the efficacy and safety of epirubicin combined with taxanes chemotherapy in the treatment of 48 cases of breast cancer in high altitude areas of Tibet. It was found that 89.5% of the patients with neutropenia after chemotherapy were significantly higher than those in low altitude areas, which also confirmed this phenomenon. The increased side effects of chemotherapy and radiotherapy in cancer patients at high altitude are closely related to hypoxia. The oxygen content and oxygen partial pressure in the atmosphere of plateau area also decrease with the increase of altitude, and the oxygen partial pressure in human alveoli also decreases, so the arterial oxygen partial pressure and saturation also decrease. A number of studies have shown that the special hypoxia environment at high altitude will have a lot of effects on the human body. In terms of cardiovascular system, it will make pulmonary hypertension and heart rate increase, and make the heart bear a heavy pressure load, leading to the occurrence of high altitude heart disease. In terms of nervous system, chronic hypoxia environment is prone to sleep disordered breathing at night, which seriously affects the brain nerve function and leads to heart failure sleep structure disorder. On the other hand, in order to adapt to the outside world, the human body in the plateau environment, within a certain limit, through the regulation of the nervous system and body fluid mechanism, carries out a series of adjustments and stress reactions, It makes a series of physiological changes in body fluid, hemorheology, blood biochemistry, blood gas and organ function, and some pathological changes, resulting in changes in physiological indexes, drug plasma protein binding rate, drug metabolic enzyme activity and expression, and inflammatory factors in blood. The investigators speculate that the above factors lead to the increase of side effects after chemotherapy at high altitude, especially the influence of inflammatory cytokines in the blood, leading to the occurrence of CRF.

ELIGIBILITY:
Inclusion Criteria:

1. Female breast cancer patients aged ≥ 18 years old;
2. Breast cancer was confirmed by histopathological investigation;
3. Chemotherapy including neoadjuvant chemotherapy, postoperative adjuvant chemotherapy and palliative chemotherapy for advanced breast cancer;
4. Eastern Cooperative Oncology Group（ECOG ）score of physical condition (0-1);
5. Voluntarily participate in the clinical trial and sign the informed consent form after informed consent (patients voluntarily accept the test and give informed consent);
6. The basic indexes were consistent, and the blood routine and ECG were normal;
7. Before chemotherapy, fatigue scale was used to score, and no fatigue symptom was confirmed by CIS and BFI;

Exclusion Criteria:

1. Due to nervous system disease, difficulty in understanding and / or lack of personnel unable to complete the report;
2. The patients were treated with radiotherapy at the same time of chemotherapy; 3.There were no other tumors, and brain metastases and pleural effusion were excluded;

4.Women diagnosed with untreated anemia and thyroid dysfunction； 5.Heart and lung diseases were excluded; 6.The respiratory system diseases affecting blood oxygen saturation were excluded; 7.Fatigue symptoms were confirmed by cis and BFI.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Fatigue was measured by Checklist for Individual Strength（CIS）. | The difference of fatigue degree between the two groups on baseline and third day after chemotherapy
  We use the Checklist for Individual Strength（CIS）fatigue scale to compare the fatigue degree of the experimental group and the control group before and after chemotherapy. In our study, we selected 8 questions in the CIS scale, each patient should answer these 8 questions, and then record the score according to the patients' answers. Each question can be scored according to absolute right and absolute wrong, and the score is from 8 to 56.

SECONDARY OUTCOMES:
Fatigue was measured by Brief Fatigue Inventory (BFI) . | The difference of fatigue degree between the two groups on baseline and third day after chemotherapy
  We used the Brief Fatigue Inventory (BFI) to compare the fatigue degree of the experimental group and the control group before and after chemotherapy. There are four questions in the BFI. The fourth question contains six small questions. The score of the questionnaire ranges from 0 to 90.
Blood pressure | The day before chemotherapy and the third day after chemotherapy.
  Blood pressure refers to the lateral pressure of blood flow in blood vessels, including systolic pressure and diastolic pressure. We use mmHg to measure blood pressure.
Biomarker in blood | The difference Biomarker level between the two groups on baseline and third day after chemotherapy
  pro-inflammatory cytokines IL-1 β, IL-6, C-reactive protein (CRP) , soluble tumor necrosis factor (TNF) receptor II (sTNF-RII),transforming growth factor (TGF-β) , Hypoxia inducible factor-1(HIF-1) , Hypoxia inducible factor-2(HIF-2)
Oxygen saturation | The day before chemotherapy and the third day after chemotherapy.
  It is the percentage of oxygenated hemoglobin volume in the blood, that is, the oxygen concentration in the blood, which is called arterial oxygen saturation. It is usually measured by the percentage sign (%).
Heart rate | The day before chemotherapy and the third day after chemotherapy.
  Heart rate refers to the number of heart beats per minute in a normal person's quiet state, also known as the quiet heart rate, which is generally 60-100 beats per minute. We use beats per minute to measure it.

CONTACTS AND LOCATIONS:
Locations (1):
- Qinghai University Affiliated Hospital, Xining, Qinghai, China

IPD SHARING:
Plan to Share IPD: No